CLINICAL TRIAL: NCT03677115
Title: Thoracic Paravertebral Blocks Using a Combination of Ropivacaine and Dexmedetomidine
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Professor, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201707158
Record Dates: First submitted 2018-09-16; First posted 2018-09-19 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Thoracic Paravertebral Blocks
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: a single-dose thoracic paravertebral analgesia for postoperative pain control after thoracoscopic lobectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dexmedetomidine group (Experimental): a combination of ropivacaine and dexmedetomidine
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — combination of ropivacaine and dexmedetomidine 20 ug every time

SUMMARY:
The investigators designed a study to assess whether thoracic paravertebral blocks using a combination of ropivacaine and dexmedetomidine prolong nerve block duration.

DETAILED DESCRIPTION:
The investigators designed a study to assess whether thoracic paravertebral blocks using a combination of ropivacaine and dexmedetomidine prolong nerve block duration. The effects of dexmedetomidine have only been compared at lower doses. This trial examined the effect of greater dose of dexmedetomidine on thoracic paravertebral block analgesia duration.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included in the study if they were ethnic Chinese,
* American Society of Anesthesiologists (ASA) physical status I or II,
* candidates for general anesthesia undergoing thoracic surgery

Exclusion Criteria:

* Patients were excluded if they do not want to cooperate with the test,
* had a history of radial artery puncture or coronary artery bypass grafting,
* had acute vessel trauma,or had been diagnosed with Raynaud' disease,
* had suffered from mental or neurological disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Change of analgesia duration | Change from Baseline to 3 days after surgery
  Change of thoracic paravertebral block analgesia duration

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided